CLINICAL TRIAL: NCT06163950
Title: The Decline in Walking Performance in Adults With Cerebral Palsy - Influence of Performance Fatigability
Acronym: FAT-GAIT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of inclusion
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22CH527; 2022-A02510-43 (Other: ANSM)
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Muscle Spasticity; Paralysis; Cerebral
Keywords: Fatigue; fatigue-resistance; torque; power; Cerebral Palsy
MeSH Terms: conditions — Muscle Spasticity; Cerebral Palsy; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with cerebral palsy (Experimental): A specially adapted recumbent cycle ergometer with the ability to quickly transform into an isometric dynamometer will be used to assess fatigability development during a task to failure. Throughout the task, which consists of blocks of 3 minutes, neuromuscular assessments will take place to determine the evolution of fatigability and its peripheral and central determinants.
  Interventions: Other: Fatigability assessment
- Healthy people (Active Comparator): A specially adapted recumbent cycle ergometer with the ability to quickly transform into an isometric dynamometer will be used to assess fatigability development during a task to failure. Throughout the task, which consists of blocks of 3 minutes, neuromuscular assessments will take place to determine the evolution of fatigability and its peripheral and central determinants.
  Interventions: Other: Fatigability assessment

INTERVENTIONS:
Other: Fatigability assessment — An isometric dynamometer will be used to assess fatigability development during a task to failure. Throughout the task, which consists of blocks of 3 minutes, neuromuscular assessments will take place to determine the evolution of fatigability and its peripheral and central determinants.

SUMMARY:
Due to an early brain injury occurring in antenatal or postnatal, cerebral palsy (CP) causes alteration in motor function with posture and gait disorders. It is commonly observed motor performance degradation during adulthood, and the underlying pathophysiology remains poorly known.

DETAILED DESCRIPTION:
One of the hypotheses to explain the decline in walking capacities in adults with CP is their greater fatigability, that could be related to energy overconsumption (due to the specific biomechanical constraints of their walking pattern) and/or the occurrence of early sarcopenia affecting the compensatory muscle mechanisms commonly seen in children to compensate for architectural disorders and posture alterations. To optimize prevention and/or therapy in these patients, it is crucial to better understand the aetiology of fatigability and its role in the decline in walking performance.

ELIGIBILITY:
Inclusion Criteria:

Common for CP and healthy volunteers:

* Capable of walking for six minutes without stopping
* Capable of consenting to the tests

Specific for the CP group

* GMFCS I or II at age 18
* Spastic diplegic cerebral palsy

Exclusion Criteria:

* Counter-indications to the test procedures
* Mental retardation or intelligence quotient (IQ) below 80
* Accompanying diseases not allowing for the test setup
* Major surgeries altering performance in the last six months
* Injection of botulin altering maximal force production in the last three months
* Refusing to sign the consent form

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Neuromuscular fatigue | Week : 6
  Neuromuscular fatigue, defined as the decrease in maximal voluntary force (in % of the resting value) developed in isometric knee extension following a standardized fatigue protocol.

SECONDARY OUTCOMES:
Maximum voluntary force torque measurement of the knee flexor muscles | Week : 2
  Measurement of the (in Nm) of the knee flexor muscles in isometric and dynamic contraction.
Maximum voluntary force torque measurement of the plantar flexor | Week : 2
  Measurement of the (in Nm) of the plantar flexor in isometric and dynamic contraction.
Maximum voluntary force torque measurement of knee extensor muscles | Week : 4
  Measurement of the (in Nm) of the knee extensor muscles in isometric and dynamic contraction.
Level of voluntary activation measurement | Week : 6
  Measurement of the level of voluntary activation (in %) determined by the force increment obtained following electrical stimulation of the motor nerve during a muscle condition of maximum contraction.
Measurement of joint amplitude (in °) | Week : 6
  Evaluation of the passive muscular properties of the dominant leg, on the knee flexor muscles, and on the plantar flexor and knee extensor muscles
Measurement of passive torque (in Nm) | Week : 6
  Evaluation of the passive muscular properties of the dominant leg, on the knee flexor muscles, and on the plantar flexor and knee extensor muscles
Evaluation of neuromuscular fatigue | Week : 6
  The decrease in muscle twitch evoked by electrical nerve stimulation (in %) (peripheral fatigue)
VO2max (in mL/min/kg) | Week : 6
  Cardiorespiratory capacity will be assessed by measuring maximal oxygen consumption (VO2max (in mL/min/kg)) in an incremental cyclo-ergometer test.
The distance covered (in m) in the 6-minute walking test | Week : 6
  Quantitative walking performance will be assessed by measuring the distance covered (in m) in the 6-minute walking test
Time (in seconds) taken during the 10-meter walk test | Week : 6
  Quantitative walking performance will be assessed by measuring the time (in seconds) taken during the 10-meter walk test
Time (in s) taken in the "Get Up and Go" test | Week : 6
  Quantitative walking performance will be assessed by measuring the time (in s) taken in the "Get Up and Go" test
Walking Quality evaluation | Week : 6
  The quality of walking will be evaluated (only in CP subjects) by a Quantified Gait Analysis (QGA) allowing the measurement of spatio-temporal parameters, joint kinematics and kinetics as well as muscle activity during walking. will be evaluated (only in CP subjects) by a Quantified Gait Analysis (QGA) allowing the measurement of spatio-temporal parameters, joint kinematics and kinetics as well as muscle activity during walking.
Berg Balance Scale | Week : 6
  Postural control (or balance) will be assessed (only in CP subjects) by the Berg Balance Scale (BBS) score. This score, ranging from 0 to 56, is an index to measure functional balance.
  0 means high risk of falling; person needs a wheelchair 56 means no risk of falling; the person has functional balance

CONTACTS AND LOCATIONS:
Overall Officials: Bruno FERNANDEZ, MD, Principal Investigator — CHU DE SAINT-ETIENNE
Locations (1):
- Centre Hospitalier de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gravholt A, Fernandez B, Rimaud D, Zeghoudi N, Bessaguet H, Espeit L, Feasson L, Millet GY, Buizer AI, Lapole T. Unravelling age-related gait decline in cerebral palsy: insights into physiological changes and functional implications through an observational study-a French study protocol in a laboratory setting. BMJ Open. 2024 Nov 27;14(11):e090096. doi: 10.1136/bmjopen-2024-090096. PMID 39609007